CLINICAL TRIAL: NCT06501625
Title: A Phase 1b/2, Safety Lead-in and Dose-Expansion, Open Label, Multicenter Trial Investigating the Safety, Tolerability, and Preliminary Activity of Ivosidenib in Combination With Durvalumab and Gemcitabine/Cisplatin as First-line Therapy in Participants With Locally Advanced, Unresectable or Metastatic Cholangiocarcinoma With an IDH1 Mutation
Brief Title: Ivosidenib Plus Durvalumab and Gemcitabine/Cisplatin as First-Line Therapy in Participants With Locally Advanced or Metastatic Cholangiocarcinoma With an IDH1 Mutation
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: S095031-210; 2024-514261-19-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-09; First posted 2024-07-15 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced, Unresectable or Metastatic Cholangiocarcinoma With an IDH1 Mutation
MeSH Terms: interventions — ivosidenib; durvalumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Safety Lead-In Phase (Experimental)
  Interventions: Drug: Ivosidenib; Drug: Durvalumab (for the first 8, 21-day, cycles); Drug: Gemcitabine (for the first 8, 21-day, cycles); Drug: Cisplatin (for the first 8, 21-day, cycles); Drug: Durvalumab (starting from cycle 9)
- Expansion Phase (Experimental)
  Interventions: Drug: Durvalumab (for the first 8, 21-day, cycles); Drug: Gemcitabine (for the first 8, 21-day, cycles); Drug: Cisplatin (for the first 8, 21-day, cycles); Drug: Durvalumab (starting from cycle 9); Drug: Ivosidenib Recommended Combination Dose (RCD)

INTERVENTIONS:
Drug: Ivosidenib — Two 250 mg tablets, totaling 500 mg, administered orally once daily, taken continuously throughout treatment duration
  Arms: Safety Lead-In Phase
Drug: Durvalumab (for the first 8, 21-day, cycles) — 1500mg intravenous (IV) infusion every 3 weeks, for a maximum of 8 (21-day) cycles
Drug: Gemcitabine (for the first 8, 21-day, cycles) — 1000 mg/m2 IV infusion on days 1 and 8 of every 21-day cycle, for a maximum of 8 cycles
Drug: Cisplatin (for the first 8, 21-day, cycles) — 25 mg/m^2 IV infusion on days 1 and 8 of every 21-day cycle, for a maximum of 8 cycles
Drug: Durvalumab (starting from cycle 9) — 1500mg intravenous (IV) infusion every 4 weeks, starting from cycle 9. Cycles are 28 days long, starting Cycle 9.
Drug: Ivosidenib Recommended Combination Dose (RCD) — RCD administered orally once daily, taken continuously throughout treatment duration
  Arms: Expansion Phase

SUMMARY:
The objective of this study is to investigate the safety, tolerability and preliminary activity of ivosidenib in combination with durvalumab and gemcitabine/cisplatin as first-line therapy in participants with locally advanced, unresectable or metastatic cholangiocarcinoma with an IDH1 mutation. The study will begin with a safety lead-in phase (Phase 1b study) to determine the recommended combination dose (RDC) and then will transition to an expansion phase (Phase 2 study) to assess the clinical activity of ivosidenib in combination with durvalumab and gemcitabine/cisplatin at the RCD. During the treatment period participants will have study visits on days 1, 8, and 15 of Cycle 1, on days 1 and 8 of Cycle 2 to 8, and on day 1 of each additional cycle. Cycles 1 through 8 are 21 day cycles, and each following cycle is 28 days. Approximately 30 days and 90 days after treatment has ended, safety follow-up visits will occur and then participants will be followed for survival every 3 months. Study visits may include blood tests, ECG, vital signs, and a physical examination.

ELIGIBILITY:
Inclusion Criteria:

* Have a histopathological confirmed diagnosis consistent with locally advanced unresectable or metastatic cholangiocarcinoma.
* Have documented IDH1 gene-mutated cholangiocarcinoma based on local or central laboratory testing (R132C/L/G/H/S mutation variants tested).
* Have at least one evaluable and measurable lesion as defined by RECIST v1.1.
* Have adequate bone marrow function as evidenced by:
* Absolute neutrophil count ≥ 1,500/mm3 or 1.5 ×109/L
* Hemoglobin ≥ 9 g/dL
* Platelet count ≥ 100,000/mm3 or 100 × 109/L
* Have adequate hepatic function as evidenced by:
* Serum bilirubin ≤ 2.0 × the upper limit of normal (ULN); this will not apply to patients with confirmed Gilbert's syndrome. Any clinically significant biliary obstruction should be resolved before randomization
* Aspartate aminotransferase (AST), and alanine aminotransferase (ALT) ≤ 2.5 × ULN; for patients with hepatic metastases, ALT and AST ≤ 5.0 × ULN
* Have adequate renal function, defined as: creatinine clearance > 60 mL/min per 24 hour urine or as calculated on the Cockcroft-Gault formula (using actual body weight):

Creatine CL (mL/min)= (140 - Age) × (weight in kg) × (0.85 if female)/72 × serum creatinine (mg/dL)

Exclusion Criteria:

* Received treatment for locally advanced, unresectable or metastatic disease with the following exceptions:
* Treatment with up to one cycle of durvalumab plus gemcitabine/cisplatin treatment is permitted before study participation. Note: For the Safety Lead-In Phase, participants who received one prior cycle of durvalumab plus gemcitabine/cisplatin and required dose modifications for treatment-related toxicity are excluded.
* Patients who developed recurrent disease > 6 months after surgery with curative intent, and, if given, > 6 months after the completion of adjuvant (chemotherapy and/or radiation).
* Prior exposure to immune-mediated therapy, including, but not limited to, anti-PD-1or other anti-PD-L1, and anti-PD-L2, anti-CTLA-4 antibodies, excluding therapeutic anticancer vaccines.
* Unresolved Grade ≥2 adverse events from a previous anticancer therapy, with the exception of alopecia and vitiligo and the laboratory values listed in the inclusion criteria.
* Patients with Grade ≥2 neuropathy to be evaluated on a case-by-case basis after consultation with the medical monitor
* Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with ivosidenib may be included only after consultation with the medical monitor
* Participation in another interventional study at the same time or within 14 days prior to the first study medication (triple combination treatment) administration. For patients having participated to another prior interventional study, the first dose of ivosidenib should occur after a period greater than or equal to 5 half-lives or 28 days, whichever is shorter of the last dose of the prior investigational product.
* Active or prior documented autoimmune or inflammatory disorders including:
* inflammatory bowel disease (e.g., colitis or Crohn's disease)
* diverticulitis (with the exception of diverticulosis)
* systemic lupus erythematosus
* Sarcoidosis syndrome
* Wegener syndrome (granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.)

Note: in cases with no active disease for ≥ 5 years, patients may be considered for inclusion if approved by the Medical Monitor. Participants with the following conditions are eligible for the study:

* chronic skin condition that does not require systemic therapy
* vitiligo
* alopecia
* hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement therapy
* unmedicated celiac disease that is controlled by diet
* Have heart rate-corrected QT interval using Fridericia's formula (QTcF) of ≥ 450 msec or with other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome/sudden death, polymorphic ventricular arrhythmia). The Sponsor should review participants with bundle branch block and prolonged QTcF for potential inclusion.
* Have an active infection, including:
* Hepatitis B (clinical evaluation includes: presence of hepatitis B surface antigen [HBsAg] and/or anti-HBcAb with detectable hepatitis B virus [HBV] DNA ≥ 10 IU/mL)
* Hepatitis C
* Tuberculosis (clinical evaluation includes: clinical history, physical examination and/or radiographic findings, and tuberculosis testing as per local practice)
* Human immunodeficiency virus (clinical evaluation includes: positive HIV 1/2 antibodies) Note: Patients with a resolved or past HBV infection (i.e., presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) do not need to be excluded from the study. Patients positive for hepatitis C (HCV) antibody are eligible only if the polymerase chain reaction is negative for HCV RNA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-07-23 (Estimated); Study Completion 2027-09-13 (Estimated)

PRIMARY OUTCOMES:
Safety Lead-in Phase: Number of Dose-limiting toxicities (DLTs) | Through Cycle 1 (Cycle 1 is 21 days)
Safety Lead-in Phase: Number of adverse events (AEs), adverse events of special interest (AESIs), and serious adverse events (SAEs) | Through 90 days after the end of treatment (Approximately 5 years)
Expansion Phase: Objective response rate (ORR) | Through the end of the study (Approximately 5 years)
  Confirmed complete response (CR) or confirmed partial response (PR) using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Safety Lead-in Phase: Ivosidenib Area under the concentration-versus-time curve (AUC) from time 0 to time of last measurable concentration (AUC0-t) | Through the end of treatment (Approximately 5 years)
Safety Lead-in Phase: Ivosidenib AUC over 1 dosing interval at steady state (AUCtau,ss) | Through the end of treatment (Approximately 5 years)
Safety Lead-in Phase: Ivosidenib time to maximum concentration (Tmax) | Through the end of treatment (Approximately 5 years)
Safety Lead-in Phase: Ivosidenib maximum concentration (Cmax) | Through the end of treatment (Approximately 5 years)
Safety Lead-in Phase: Ivosidenib trough concentration (Ctrough) | Through the end of treatment (Approximately 5 years)
Safety Lead-in Phase: Ivosidenib apparent volume of distribution (Vd/F) | Through the end of treatment (Approximately 5 years)
Safety Lead-in Phase: Ivosidenib apparent clearance (CL/F) | Through the end of treatment (Approximately 5 years)
Safety Lead-in Phase: Plasma 2-hydroxygluturate (2-HG) concentrations | Through the end of treatment (Approximately 5 years)
Expansion Phase: Number of AEs, AESIs, and SAEs | Through 90 days after the end of treatment (Approximately 5 years)
Expansion Phase: Overall survival (OS) | Through the end of the study (Approximately 5 years)
Expansion Phase: Duration of response (DOR) | Through the end of the study (Approximately 5 years)
Expansion Phase: Progression-free survival (PFS) | Through the end of the study (Approximately 5 years)
Expansion Phase: Disease control | Through the end of the study (Approximately 5 years)
  Confirmed CR, confirmed PR, or stable disease [SD]
Expansion Phase: Time to response (TTR) | Through the end of the study (Approximately 5 years)
Expansion Phase: Ivosidenib Area under the concentration-versus-time curve (AUC) from time 0 to time of last measurable concentration (AUC0-t) | Through the end of treatment (Approximately 5 years)
Expansion Phase: Ivosidenib AUC over 1 dosing interval at steady state (AUCtau,ss) | Through the end of treatment (Approximately 5 years)
Expansion Phase: Ivosidenib time to maximum concentration (Tmax) | Through the end of treatment (Approximately 5 years)
Expansion Phase: Ivosidenib maximum concentration (Cmax) | Through the end of treatment (Approximately 5 years)
Expansion Phase: Ivosidenib trough concentration (Ctrough) | Through the end of treatment (Approximately 5 years)
Expansion Phase: Ivosidenib apparent volume of distribution (Vd/F) | Through the end of treatment (Approximately 5 years)
Expansion Phase: Ivosidenib apparent clearance (CL/F) | Through the end of treatment (Approximately 5 years)
Expansion Phase: Plasma 2-hydroxygluturate (2-HG) concentrations | Through the end of treatment (Approximately 5 years)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (7):
  - Usc Norris Comprehensive Cancer Center, Los Angeles, California
  - Northwestern Medicine, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University, Durham, North Carolina
  - Gibbs Cancer Center, Spartanburg, South Carolina
  - Tennesse Oncology - Elliston Place Plaza, Nashville, Tennessee
  - The University of Texas Md Anderson Cancer Center, Houston, Texas
- Alfred Health, Melbourne, Australia
- Brazil (4):
  - Hospital de Amor - Barretos, Barretos
  - Oncoclinicas Mg, Belo Horizonte
  - CIONC, Curitiba
  - Instituto Dor de Pesquisa E Ensino Sp, São Paulo
- Princess Margaret Cancer Centre, Toronto, Canada
- France (3):
  - Institut Bergonie, Bordeaux
  - Hôpital Beaujon, Clichy
  - Chu Montpellier-Hopital Saint-Eloi, Montpellier
- Germany (5):
  - Charite Universitatsmedizin, Berlin
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitären Centrums Für Tumorerkrankungen (Uct) Der J.W. Goethe-Universität Frankfurt, Frankfurt
  - Medizinische Hochschule Hannover Oe 6810, Hanover
  - Universitätsklinikum Ulm, Ulm
- Japan (4):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Cancer Center Hospital, Chūōku
  - Kyoto University Hospital, Kyoto
  - Kanagawa Cancer Center, Yokohama
- South Korea (7):
  - Cha Bundang Medical Center, Seongnam
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance, Seoul
  - Seoul St. Mary'S Hospital, Seoul
- Spain (5):
  - H. Valle de Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Gregorio Marañón, Madrid
  - H. 12 de Octubre, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data. Access can be requested for all interventional clinical studies:
  * Used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorization in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com/